CLINICAL TRIAL: NCT00265512
Title: Improving Longterm SUD Outcomes With Telephone Case Monitoring
Brief Title: LINK: Aftercare Monitoring Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 05-021
Record Dates: First submitted 2005-12-12; First posted 2005-12-14 (Estimated); Results first posted 2014-10-17 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2018-07

CONDITIONS: Alcohol Dependence; Drug Dependence
Keywords: Telemedicine; Aftercare
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telephone Case Monitoring Aftercare (Active Comparator): Telephone Case Monitoring Aftercare
  Interventions: Behavioral: Telephone Case Monitoring
- Continuing Care as Usual (Active Comparator): Continuing Care as Usual
  Interventions: Behavioral: Continuing Care as Usual

INTERVENTIONS:
Behavioral: Telephone Case Monitoring — Telephone Case Monitoring involves telephone delivery of continuing care treatment post intensive outpatient SUD treatment. It includes brief weekly phone calls with a counselor for up to 6 months.
  Other Names: TCM
  Arms: Telephone Case Monitoring Aftercare
Behavioral: Continuing Care as Usual — Continuing Care as Usual will include standard group outpatient SUD treatment.
  Other Names: CCAU
  Arms: Continuing Care as Usual

SUMMARY:
The prevalence of substance use disorders (SUD) in the VA is rising, making SUD(s) among the most commonly diagnosed disorders in the VA. A substantial body of data attests to the effectiveness of substance use disorder treatment; further the predictor most consistently associated with positive addiction treatment outcomes is duration. Despite the body of evidence supporting length of treatment as one of the stronger predictors of long-term SUD outcomes, only 36% of SUD treatment programs in the VA are meeting the continuing care performance criterion specified by the Office of Quality Performance. This randomized clinical trial investigates whether substance use disorder patients assigned to telephone case monitoring (TCM) for continuing care will do better than those attending face-to-face continuing care as usual (CCAU)(standard outpatient care).

DETAILED DESCRIPTION:
Background: The prevalence of substance use disorders (SUD) in the VA is rising, making SUD(s) among the most commonly diagnosed disorders in the VA. A substantial body of data attests to the effectiveness of substance use disorder treatment; further the predictor most consistently associated with positive addiction treatment outcomes is duration. Despite the body of evidence supporting length of treatment as one of the stronger predictors of long-term SUD outcomes, only 36% of SUD treatment programs in the VA are meeting the continuing care performance criterion specified by the Office of Quality Performance. The proposed randomized clinical trial investigates whether substance use disorder patients assigned to telephone case monitoring (TCM) for continuing care will do better than those attending face-to-face continuing care as usual (CCAU)(standard outpatient care).

Objectives: The objective of this research is to test, in a randomized clinical trial, whether in-person CCAU following intensive outpatient SUD treatment leads to better SUD outcomes when compared with TCM. In addition, we will investigate whether continuing care condition interacts with distance from providers such that telephone case monitoring (TCM) produces increasingly stronger results relative to continuing care as usual (CCAU) as distance from care increases. Should we find an interaction, we will test whether the interaction is due to TCM producing better proximal outcomes such as level of participation in continuing care and satisfaction with treatment. Finally, we will investigate the cost of providing telephone care relative to continuing care as usual.

Methods: The design of this study is a randomized controlled trial of telephone case monitoring versus face-to-face continuing care as usual with 2 sites and up to 500 patients per site recruited over 1.5 years for a total of up to 1000 patients. Patients will be involved in the intervention for up to 6 months and data collection will occur at baseline, 3, 6 and 12 months via mailed surveys. Data of interest include self-report of substance use, psychiatric symptoms, and quality of life. Data analyses will be conducted using hierarchical linear modeling.

Status: Patient recruitment has ended. Treatment and follow-up are on-going.

ELIGIBILITY:
Inclusion Criteria:

Participants will be recruited from all patients who complete at least 14 days of intensive outpatient (IOP) substance use disorder treatment over an 18-month period in 2 VA IOP SUD programs.

Exclusion Criteria:

Completion of less than 14 days of IOP treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 667 (Actual)
Dates: Start 2006-11; Primary Completion 2009-06 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D. McKellar, PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (3):
- United States (3):
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA Eastern Kansas Health Care System Colmery-O'Neil VA Medical Center, Topeka, KS, Topeka, Kansas
  - St. Louis VA Medical Center John Cochran Division, St. Louis, MO, St Louis, Missouri

REFERENCES:
- [Result] McKellar J, Wagner T, Harris A, Oehlert M, Buckley S, Moos R. One-year outcomes of telephone case monitoring for patients with substance use disorder. Addict Behav. 2012 Oct;37(10):1069-74. doi: 10.1016/j.addbeh.2012.03.009. Epub 2012 Mar 13. PMID 22651986
- [Result] Oser M, Cucciare M, McKellar J, Weingardt K. Correlates of hazardous drinking among Veterans with and without hepatitis C. J Behav Med. 2012 Dec;35(6):634-41. doi: 10.1007/s10865-011-9394-9. Epub 2012 Jan 11. PMID 22234384
- [Result] Austin J, McKellar JD, Moos R. The influence of co-occurring axis I disorders on treatment utilization and outcome in homeless patients with substance use disorders. Addict Behav. 2011 Sep;36(9):941-4. doi: 10.1016/j.addbeh.2011.05.001. Epub 2011 May 7. PMID 21620571
- [Result] Oser ML, McKellar J, Moos BS, Moos RH. Changes in ambivalence mediate the relation between entering treatment and change in alcohol use and problems. Addict Behav. 2010 Apr;35(4):367-9. doi: 10.1016/j.addbeh.2009.10.024. Epub 2009 Oct 30. PMID 19926399
- [Result] Barbosa PV, Thomas IC, Srinivas S, Buyyounouski MK, Chung BI, Chertow GM, Asch SM, Wagner TH, Brooks JD, Leppert JT. Overall Survival in Patients with Localized Prostate Cancer in the US Veterans Health Administration: Is PIVOT Generalizable? Eur Urol. 2016 Aug;70(2):227-30. doi: 10.1016/j.eururo.2016.02.037. Epub 2016 Mar 2. PMID 26948397
- [Result] Wagner TH, Burstin H, Frakt AB, Krein SL, Lorenz K, Maciejewski ML, Pizer SD, Weiner M, Yoon J, Zulman DM, Asch SM. Opportunities to Enhance Value-Related Research in the U.S. Department of Veterans Affairs. J Gen Intern Med. 2016 Apr;31 Suppl 1(Suppl 1):78-83. doi: 10.1007/s11606-015-3538-5. No abstract available. PMID 26951279
- [Result] Gidwani R, Joyce N, Kinosian B, Faricy-Anderson K, Levy C, Miller SC, Ersek M, Wagner T, Mor V. Gap between Recommendations and Practice of Palliative Care and Hospice in Cancer Patients. J Palliat Med. 2016 Sep;19(9):957-63. doi: 10.1089/jpm.2015.0514. Epub 2016 May 26. PMID 27228478

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Telephone Case Monitoring Aftercare | Continuing Care as Usual
Started | 213 | 454
Completed | 168 | 359
Not Completed | 45 | 95

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telephone Case Monitoring Aftercare | Continuing Care as Usual | Total
Number analyzed (Participants) | 213 | 454 | 667
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (8.5) | 51.0 (8.1) | 51.3 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 21 | 31
  Male | 203 | 433 | 636

OUTCOME MEASURES:

1. Primary Outcome: Rates of Substance Use
Description: Percentage of days abstinent from alcohol use. Each person is followed for 3 months. For each person, we then calculate the number of days they were abstinent and the percentage of days abstinent (days abstinent/ all days in 3 months).
Time Frame: Rates of substance use measured at 3 months
Measure: Mean (Standard Error); unit: percentage of days
Arm/Group | Telephone Case Monitoring Aftercare | Continuing Care as Usual
Number analyzed (Participants) | 213 | 454
percentage of days | 91.1 (1.79) | 88.0 (1.81)

2. Secondary Outcome: Psychiatric Symptoms
Description: 3 month, 6 month and 12 month measures of psychiatric symptoms, as measured by the Brief Symptom Inventory (BSI). Minimum observed score was 22; maximum observed score was 110. Higher score is worse. Minimum score possible is 22. Maximum score possible is 110.
Time Frame: Psychiatric symptoms measured at 3 months, 6 months, 12 months post randomization
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Telephone Case Monitoring Aftercare | Continuing Care as Usual
Number analyzed (Participants) | 213 | 454
score on a scale
  3 months | 47.22 (1.41) | 50.50 (1.00)
  6 months | 49.76 (1.42) | 51.88 (1.02)
  12 months | 48.79 (1.47) | 51.18 (1.07)

3. Secondary Outcome: Health Related Quality of Life
Description: Physical and mental health subscales from the 12-item Medical Outcomes Study Short-form Health Survey, adapted for Veterans (VR-12). Observed scores on the MCS ranged from 2.89 to 70.39. Scores on the PCS ranged from 13.26 to 70.10. Higher scores denote better health. The minimum and maximum scores possible are 0 and 100, respectively.
Time Frame: 3 months, 6 months and 12 months after randomization
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Telephone Case Monitoring Aftercare | Continuing Care as Usual
Number analyzed (Participants) | 209 | 443
score on a scale
  3 month PCS | 45.64 (.83) | 44.92 (.57)
  6 month PCS | 44.54 (.96) | 43.58 (.66)
  12 month PCS | 43.37 (.91) | 42.72 (.66)
  3 month MCS | 36.22 (.81) | 35.13 (.57)
  6 month MCS | 40.81 (1.02) | 39.09 (.66)
  12 month MCS | 40.72 (.94) | 40.12 (.69)

ADVERSE EVENTS:
Description: Serious Adverse Events were tracked. There was no tracking of other adverse events.
Groups:
- Telephone Case Monitoring Aftercare: Telephone Case Monitoring: Telephone Case Monitoring involves telephone delivery of continuing care treatment post intensive outpatient SUD treatment. It includes brief weekly phone calls with a counselor for up to 6 months.
  SAEs were tracked, but AEs were not tracked.
- Continuing Care as Usual: Continuing Care as Usual: Continuing Care as Usual will include standard group outpatient SUD treatment.
  SAEs were tracked, but AEs were not tracked.
Arm/Group | Telephone Case Monitoring Aftercare | Continuing Care as Usual
All-Cause Mortality (participants affected / at risk) | 0/213 | 0/454
Serious Adverse Events (participants affected / at risk) | 60/213 | 92/454
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telephone Case Monitoring Aftercare (N=213) | Continuing Care as Usual (N=454)
hosapitalizations (General disorders) | 60 (102) | 92 (206)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No